CLINICAL TRIAL: NCT02062892
Title: Differentiating Sirolimus and Everolimus in Combination With Calcineurin Inhibitors in Long-term Maintenance of Kidney Transplant Patients - The Effects on Vascular Endothelial and Kidney Function. The DESIRE Study.
Brief Title: Differentiating Everolimus Versus Sirolimus in Combination With Calcineurin Inhibitors in Kidney Transplant Patients
Acronym: DESIRE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients meeting the inclusion/ exclusion criteria did not agree to participate. It became obvious that recruitment goals could not be met.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 13-1583; CRAD001AUS196T (Other)
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Transplantation
Keywords: everolimus; sirolimus; tacrolimus; vascular endothelial function; kidney; Transplantation; biomarkers
MeSH Terms: interventions — Everolimus; Sirolimus

ARMS (2):
- Everolimus / Tacrolimus (Experimental): Patients will be stable kidney transplant patients who are receiving an immunosuppressive drug regimen based on tacrolimus and sirolimus. 24 hours after the last sirolimus dose, the patients randomized to the tacrolimus/everolimus arm of the study will be switched from sirolimus to everolimus 1:1 (same sirolimus as everolimus dose). Everolimus doses will be adjusted so that trough blood concentrations are within 3-8 ng/mL. In detail: Tacrolimus (Prograf or FDA approved generic 0.5 mg, 1 mg or 5 mg capsules, twice a day) in combination with Everolimus (Zortress, 0.25, 0.5 and 0.75 tablets).
  Interventions: Drug: Everolimus
- Sirolimus / Tacrolimus (Active Comparator): Patients will be stable kidney transplant patients who are receiving an immunosuppressive drug regimen based on tacrolimus and sirolimus. 24 hours after the last sirolimus dose, the patients randomized to the tacrolimus/sirolimus arm of the study will remain on tacrolimus/sirolimus. In detail: Tacrolimus (Prograf or FDA approved generic 0.5 mg, 1 mg or 5 mg capsules, once a day) in combination with Sirolimus (Rapamune, 0.5, 1, and 2mg tablets).
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Everolimus — Patients will be stable kidney transplant patients who are receiving an immunosuppressive drug regimen based on tacrolimus and sirolimus. 24 hours after the last sirolimus dose, the patients randomized to the tacrolimus/everolimus arm of the study will be switched from sirolimus to everolimus 1:1 (same sirolimus as everolimus dose). Everolimus doses will be adjusted so that trough blood concentrations are within 3-8 ng/mL. In detail: Tacrolimus (Prograf or FDA approved generic 0.5 mg, 1 mg or 5 mg capsules, twice a day) in combination with Everolimus (Zortress, 0.25, 0.5 and 0.75 tablets).
  Other Names: Zortress
  Arms: Everolimus / Tacrolimus
Drug: Sirolimus — Patients will be stable kidney transplant patients who are receiving an immunosuppressive drug regimen based on tacrolimus and sirolimus. 24 hours after the last sirolimus dose, the patients randomized to the tacrolimus/sirolimus arm of the study will remain on tacrolimus/sirolimus. In detail: Tacrolimus (Prograf or FDA approved generic 0.5 mg, 1 mg or 5 mg capsules, once a day) in combination with Sirolimus (Rapamune, 0.5, 1, and 2mg tablets).
  Arms: Sirolimus / Tacrolimus

SUMMARY:
The investigators hypothesize that switching kidney transplant patients on tacrolimus/sirolimus long-term maintenance immunosuppressive drug regimens to tacrolimus/everolimus, will not only be safe, but will lead to better kidney function than patients staying on tacrolimus/sirolimus due to the lower potential of everolimus to enhance calcineurin inhibitors toxicity and/or its ability to even reverse some of the negative effects of calcineurin inhibitors on vascular endothelial and kidney function. To test this hypothesis vascular endothelial biomarkers will be analyzed in blood plasma samples and kidney dysfunction biomarkers in urine samples via liquid chromatography tandem mass spectrometry to evaluate whether switching kidney transplant patients on tacrolimus/sirolimus to tacrolimus/everolimus will lead to better kidney and endothelial function after one year and two years.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients ≥ 3 months after transplantation. De novo patients on sirolimus and tacrolimus as well as patients switched to tacrolimus and sirolimus will be eligible as long as they have received this drug combination for at least 2 months.
* Immunosuppressive drug regimen based on tacrolimus and sirolimus
* 18-70 years of age
* calculated glomerular filtration rate≥ 30 mL/min/ 1.73m2 as calculated using the abbreviated Modification of Diet in Renal Disease formula
* Ability and willingness to provide written informed consent and adhere to study regimen.
* Patients who are able to take oral medication at time of randomization.

Exclusion Criteria:

* Patients switched to tacrolimus and sirolimus due to clinically relevant nephrotoxicity of the previous immunosuppressive drug regimen,
* Patients with an abnormal liver profile such as alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin > 3 x upper limit of normal at time of randomization
* Patients with severe total hypercholesterolemia (> 350 mg/dL; > 9 mmol/L) or total hypertriglyceridemia (> 500 mg/dL; > 5.6 mmol/L). Patients on lipid lowering treatment with controlled hyperlipidemia are acceptable.
* Patients who tested positive for HIV, Hepatitis C or Hepatitis B surface antigen.
* An episode of acute rejection that required antibody therapy or more than one steroid sensitive episode of acute rejection prior to enrollment.
* Spot urine protein/creatinine ratio > 1g/24h at the time of randomization
* Multi-organ transplants
* Patients with platelet count < 50,000
* Patients with an absolute neutrophil count of < 1,000 or white blood cells of <2,000 at time of enrollment
* Patients with hemoglobin < 6g/dL
* Patients with clinically significant systemic infections requiring active use of IV antibiotics, anti-virales, or anti-fungals. Prophylactic use of anti-virales will be acceptable.
* Pregnancy or inability of practicing acceptable contraceptive measures.
* Patients who have any surgical or medical condition, such as severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, which in the opinion of the investigator might significantly alter the absorption, distribution, metabolism and/or excretion of study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Creatinine Outcome Measure (1) | 1 year
  Kidney function outcome markers will be assessed one year after kidney transplant
Calculated Glomerular Filtration Rate (1) | 1 year
  Kidney function outcome markers will be assessed one year after kidney transplant
Calculated Glomerular Filtration Rate (2) | 2 years
  Kidney function outcome markers will be assessed two years after kidney transplant
Kidney Injury Molecule-1 (1) | 1 year
  Kidney function outcome markers will be assessed one year after kidney transplant
Kidney Injury Molecule-1 (2) | 2 years
  Kidney function outcome markers will be assessed two years after kidney transplant
S-Adenosylhomocysteine Hydrolase (1) | 1 year
  Kidney function outcome markers will be assessed one year after kidney transplant
S-Adenosylhomocysteine Hydrolase (2) | 2 years
  Kidney function outcome markers will be assessed two years after kidney transplant
S-Adenosylmethionine (1) | 1 year
  Kidney function outcome markers will be assessed one year after kidney transplant
S-Adenosylmethionine (2) | 2 years
  Kidney function outcome markers will be assessed two years after kidney transplant
Creatinine Outcome Measure (2) | 2 years
  Kidney function outcome markers will be assessed two years after kidney transplant

SECONDARY OUTCOMES:
12-Hydroxyeicosatetraenoic acid (1) | 1 year
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant
12-Hydroxyeicosatetraenoic acid (2) | 2 years
  Vascular endothelial dysfunction outcome markers will be assessed two years after kidney transplant
20-Hydroxyeicosatetraenoic acid (1) | 1 year
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant
20-Hydroxyeicosatetraenoic acid (2) | 2 years
  Vascular endothelial dysfunction outcome markers will be assessed two years after kidney transplant
18- Hydroxyeicosapentaenoic acid (1) | 1 year
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant
18- Hydroxy- eicosapentaenoic acid (2) | 2 years
  Vascular endothelial dysfunction outcome markers will be assessed two years after kidney transplant
Ornithine (1) | 1 year
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant
Ornithine (2) | 2 years
  Vascular endothelial dysfunction outcome markers will be assessed two years after kidney transplant
Arginine (1) | 1 year
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant
Arginine (2) | 2 years
  Vascular endothelial dysfunction outcome markers will be assessed one year after kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Chan, MD, PhD, Principal Investigator — University of Colorado, Denver; Clifford Miles, MD, MS, Principal Investigator — University of Nebraska